CLINICAL TRIAL: NCT04767997
Title: Effects of Probiotics on Sleep Quality Among Mildly Stressed Adults: A Randomized, Placebo-controlled, Double-blind, Parallel Trial
Brief Title: Probiotics on Sleep Among Adults Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: L-019
Record Dates: First submitted 2021-02-19; First posted 2021-02-24 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Sleep Disturbance; Sleep Patterns
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants in this group will be randomized to receive probiotic formulation for the following 12 weeks.
  Interventions: Dietary Supplement: Probiotic formulation
- Control group (Placebo Comparator): Participants in this group will be randomized to receive placebo for the following 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic formulation — Participants will be asked to take one capsule daily, containing 3 billion CFU of the probiotics.
  Arms: Experimental group
Dietary Supplement: Placebo — Participants will be asked to take a placebo capsule daily.
  Arms: Control group

SUMMARY:
The aim of this study is to determine the impact of a probiotic formulation on subjective sleep patterns. It is hypothesized that participants given the probiotics will improve their sleep patterns compared to participants receiving placebo.

DETAILED DESCRIPTION:
Participants with symptoms of insomnia and work-related stress will be recruited to participate in a randomized, placebo-controlled, double-blind interventional study for approximately 15 since the signature of the informed consent. Participants will first be seen at the Screening visit when they will be administered several questionnaires to determine eligibility (assessing symptoms of insomnia, work-related stress, psychological distress and other sleep disorders). Participants will receive a 2-week sleep journal and an actigraphy to record their sleep patterns. At visit 2 returning participants will be randomized to receive probiotics or placebo for the following 12 weeks. During this visit, participants will be administered questionnaires assessing sleep quality, work-related productivity, quality of life, and mood. Participants will also be asked to bring to site a stool sample and saliva samples.

Participants will be asked to return at 6 weeks for visit 3. During this visit participants will be administered questionnaires (insomnia, sleep quality, work-related stress and productivity, quality of life, mood and psychological distress).

They will also bring two saliva samples. Two weeks prior to visit 4, participants will be asked to complete another sleep journal and be dispensed another actigraphy which shall be returned at visit 4. Lastly, participants will return on for visit 4 at week 12 in which the same questionnaires as visit 3 will be administered. Participants will also be asked to bring to site another stool sample and two saliva samples.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged between 18 and 65 years-old
2. Scores 8 ≥ in the ISI
3. Having a score higher to 0.8 in the ERI questionnaire
4. Body mass index (BMI) below or equal to 30.
5. Otherwise healthy
6. Working (paid or unpaid) at the same position for at least the past 3 months and plans to have the same position for the duration of the study.
7. Willing to discontinue consumption of probiotics supplements and probiotic fortified products throughout the study

Exclusion Criteria:

1. Presence of unrelated sleep disorders (Obstructive Sleep Apnea and REM Sleep Behavior Disorder) as per questionnaires (STOP BANG and the RBD single question, respectively).
2. Diagnosis of mental disorders (diagnosed by a health professional in the last year, including insomnia) or showing high psychosocial stress assessed by K10 (score equal or above 17).
3. Diabetes (type I and II), blood/bleeding disorders, liver and/or kidney disorders, unstable cardiovascular diseases, neurological diseases (such as, but not limited to Alzheimer's disease, Parkinson's disease, epilepsy), gastrointestinal diseases (such as, but not limited to gastric ulcers, Crohn's disease, ulcerative colitis).
4. Irregular bedtime schedule (schedule resulting in usual bedtime earlier than 8 PM or later than 2 AM or arising time earlier than 4 AM or later than 10 AM).
5. Currently suffering from periodontitis.
6. Pregnancy, planning to be pregnant or currently breastfeeding.
7. Use of medication to improve sleep, such as Zopiclone, Doxepine, Trazodone, Melatonin, any H1-antagonist, antipsychotics.
8. Milk and soy allergy.
9. Lactose intolerance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Symptoms of insomnia | 12 weeks
  Comparison of sleep quality assessed by the Insomnia Severity Index among probiotic versus placebo

SECONDARY OUTCOMES:
Symptoms of insomnia (progressive treatment) | 6 weeks
  Comparison of sleep quality assessed by the Insomnia Severity Index among probiotics versus placebo
Objective assessment of sleep: Sleep Latency | 12 weeks
  Comparison of sleep latency recorded by actigraphy of probiotic versus placebo
Objective assessment of sleep: Sleep Efficiency | 12 weeks
  Comparison of sleep efficiency recorded by actigraphy of probiotic versus placebo
Objective assessment of sleep: Wake after sleep onset (WASO) | 12 weeks
  Comparison of WASO recorded by actigraphy of probiotic versus placebo
Subjective sleep patterns | 12 weeks
  Comparison of sleep quality, assessed via Visual Analogue Scale (0 to 12; higher scores indicate worse sleep patterns), among probiotics versus placebo
Subjective sleep patterns (progressive treatment) | 6 weeks
  Comparison of sleep quality, assessed via Visual Analogue Scale (0 to 12; higher scores indicate worse sleep patterns), among probiotics versus placebo
Work-related stress | 12 weeks
  Comparison of overall score obtained at the Effort-Reward Imbalance (ERI; scores below 0.8 denote higher reward) among probiotics versus placebo
Work Productivity | 12 weeks
  Comparison of overall score obtained at the Work Productivity and Activity Impairment (WPAI; 0% to 100%, with higher scores indicating higher impairment and lower productivity) questionnaire among probiotics versus placebo groups.
Change on Quality of life | 12 weeks
  Comparison of overall score obtained at the questionnaires WHOQOL-Bref (0 to 100; higher scores denote higher quality of life) and Kessler 10 (K10; 5 - no psychological distress to 50 - high psychological distress) among probiotics versus placebo groups.
Mood | 12 weeks
  Comparison of overall score obtained at the HADS questionnaire (0 - no mood disorder to 21 - responder likely suffers depression and/or anxiety) among probiotics versus placebo groups.
Levels of sleep-related hormones | 12 weeks
  Comparison of the cortisol and melatonin quantified from saliva samples among probiotics versus placebo
Safety of intervention (number of Serious and Adverse events) | 12 weeks
  Comparison of the number of adverse events and serious adverse events reported by participants randomized to receive probiotics compared to those receiving placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Morin, Ph.D., Principal Investigator — Centre de recherche CERVO
Locations (1):
- Centre d'étude des troubles du sommeil, Centre de recherche CERVO/BRAIN, Québec, Canada

IPD SHARING:
Plan to Share IPD: No
After publications of the results, de-identified data will be shared with qualified researchers and scientists upon reasonable request to the sponsor including a detailed proposal of the intended use of the data, as per the Lallemand Health Solutions Inc. Policy on Clinical Trial Transparency and Data Sharing (available upon request).